CLINICAL TRIAL: NCT03148990
Title: A Phase II / III, Clinical Trial to Evaluate the Immunogenicity, Reatogenicity and Safety of Double Viral Vaccine (MR) for Measles and Rubella, Produced by Bio-Manguinhos / Fiocruz in 11-month-old Infants.
Brief Title: Study to Evaluate the Immunogenicity, Reatogenicity and Safety of Double Viral Vaccine (MR) for Measles and Rubella
Acronym: BIOMR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Oswaldo Cruz Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ASCLIN 002/2017
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2019-05

CONDITIONS: Rubella; Measles
Keywords: Double Viral Vaccine Measles and Rubella; Safety Efficacy Imunogenicity
MeSH Terms: conditions — Rubella; Measles | interventions — Rubella Vaccine; Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Intervention Model Description: Two intervention groups (MR vaccine and MMR vaccine), with 1 dose of vaccine in each group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measles and Rubella vaccine (Experimental): Biological/Vaccine: Administration of the experimental vaccine (Measles and Rubella).
  Interventions: Biological: Measles and Rubella vaccine
- Measles, Mumps and Rubella vaccine (Active Comparator): Biological/Vaccine: Administration of the comparator vaccine (Measles, Mumps and Rubella).
  Interventions: Biological: Measles, Mumps and Rubella vaccine

INTERVENTIONS:
Biological: Measles and Rubella vaccine — Administration of the experimental vaccine (MR).
  Arms: Measles and Rubella vaccine
Biological: Measles, Mumps and Rubella vaccine — Administration of the comparator vaccine (MMR).
  Arms: Measles, Mumps and Rubella vaccine

SUMMARY:
Measles and rubella are highly contagious acute viral diseases. As per WHO, several evidences demonstrate the benefit for providing the universal access to vaccines containing measles and rubella antigens, mainly due to, respectively, mortality in children and malformations in fetuses. This is a Phase I-III, Controlled, randomized and double blind for the evaluation double viral vaccine anti-measles and rubella (MR), which is developed and produced at Instituto de Tecnologia em Imunobiologicos Bio-Manguinhos/Fiocruz, in Brazil, for use in human beings. 432 eligible volunteers (11-month-old infants), will be vaccinated and monitored for local and systemic adverse events and titration of antibodies. The study will last 11 months in total.

DETAILED DESCRIPTION:
This is a Phase II-III, controlled, randomized and double blind for the evaluation of a double viral vaccine anti measles and rubella (MR), which is under the development at Instituto de Tecnologia em Imunobiologicos Bio-Manguinhos/Fiocruz, in Brazil, for use in human beings. 432 eligible volunteers (11-month-old infants), will be vaccinated and monitored for local and systemic adverse events and immunogenicity. The study will last 11 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Both sex;
* Good health (no significant medical history);
* 11 months of age on the first dose of vaccine;
* To be up-to-date with the national vaccination calendar;
* Availability for follow-up throughout the study period;
* Willing to provide name, address, telephone and other contact information in order to be contacted, whenever needed (example: in case of missing any scheduled visit, contact for confirmation of scheduling a visit, urgent safety notifications);
* Willing to strictly follow the study protocol;
* At least one legal guardian of the research participants must be able to understand and sign the informed consent form;
* Legal guardians by the research participants who can understand the child's inability to participate in another clinical trial during the time they are participating in the study;
* Legal guardian with intellectual capacity to fill out the signs of signs and symptoms at home.

Exclusion Criteria:

* Previous vaccination against measles and rubella;
* Personal history of measles or rubella;
* Personal history of anaphylactic shock, asthma, urticaria or other hypersensitivity reaction to previous vaccinations, or who are allergic or hypersensitive to vaccine components of the study;
* Use of antiallergic injections with antigens within 14 days or less prior to vaccination;
* Use of immunoglobulin in the last 12 months prior to vaccination;
* Use of blood products in the last 12 months prior to vaccination;
* Use of any type of vaccine less than 30 days prior to study vaccination;
* Use of injectable vaccines less than 42 days after study vaccination;
* Chronic use of any medications (except homeopathic medicines and trivial medication such as saline and vitamins);
* Previous use of immunosuppressive or cytotoxic medication;
* Use of systemic therapy with high doses of steroids;
* Use of any type of medication in a clinical trial within 12 months prior to vaccination;
* Personal history of clinically significant neurological, cardiovascular, respiratory, hepatic, renal, haematological, rheumatologic or autoimmune diseases;
* Personal history of coagulopathies diagnosed by a physician or report of capillary fragility;
* Personal history of seizures;
* Personal history of an active (eg any cancer) or treated malignant disease that may recur during the study;
* Personal history of sickle cell anemia;
* Asplenia (absence of spleen or removal of the spleen);
* HIV positive or history of any immunosuppressive disease;
* Presence of any disorder which, in the opinion of the principal investigator, may interfere with the evaluation of the study objectives;
* Legal guardian with limited capacity for adherence to the study, according to the researcher's evaluation;
* Impossibility of blood collection for pre-vaccine evaluation.

Ages: 11 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 432 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity analysis of the study vaccine | 42 days after the 1st dose of MR or MMR
  To evaluate imune response between post and pre-vaccination antibodies.

SECONDARY OUTCOMES:
Reatogenicity analysis of the study vaccine | 30 days after the 1st dose of MR or MMR
  To assess the occurrence of serious adverse events among individuals who received MR and MMR vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Kleber G Luz, PhD, Principal Investigator — Centro de Estudos e Pesquisas em Moléstias Infecciosas Ltda
Locations (2):
- Brazil (2):
  - Centro de Estudos e Pesquisas em Moléstias Infecciosas Ltda (CPCLIN), Natal, Rio Grande do Norte
  - Secretaria Municipal de Saúde do Estado do Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No